# A Randomized Trial of Transcutaneous Nerve Stimulation for Overactive Bladder Patients

Dr Blayne Welk
Assistant Professor, Western University

NCT 02511717 March 1 2016

#### Statement of Objective

To determine the efficacy of <u>trans</u>cutaneous tibial nerve stimulation (using skin patch electrodes) for the treatment of women with clinical symptoms of overactive bladder.

#### **Background**

Overactive bladder is a clinical diagnosis characterized by "urinary urgency, often with frequency and nocturia, with or without urgency urinary incontinence"<sup>2</sup>. Approximately 16% of adult women meet the clinical definition for overactive bladder, and approximately 1/3 of them will have urgency incontinence<sup>3,4</sup>. While a small proportion of patients do see their symptoms resolve after a year, for the vast majority this is a chronic condition<sup>4,5</sup>. Although it is not inherently dangerous, overactive bladder is an important condition given its wide-ranging impact on overall quality of life and mental health<sup>3</sup>. The magnitude of impact across different domains of quality of life is similar to chronic diseases such as diabetes<sup>6</sup>. In addition, the financial impact is substantial; in the United States this has been estimated at \$12 billion annually<sup>7</sup>.

#### Hypothesis

I hypothesize that the study protocol of <u>trans</u>cutaneous tibial nerve stimulation performed at home during 30 minute sessions, 3x/week, for 12 weeks will be associated with a statistically significant improvement in overall bladder symptoms.

#### Design and methodology

Study design: This is a randomized, double blind, sham controlled clinical trial. The primary intervention is 30 minute sessions, 3x/week, for 12 weeks of transcutaneous tibial nerve stimulation sessions carried out at home. The sham intervention will consist of the same treatment schedule, except with the application of transcutaneous nerve stimulation to the lateral aspect of the lower leg, away from the tibial nerve. Patients will undergo a 12 week treatment course. The patient and the treating physician will be blinded to the group assignment of the patient. Randomization will be done using a random number generator, and study assignment will only be released at the end of the study. Only the study nurse instructing the patient on placement of the study electrodes will know the patient assignment. The effectiveness of our sham protocol will be evaluated with a question during week 2-3 asking if they think they are in the active or sham group. The study visit schedule is outlined in more detail in Appendix 2.

#### Inclusion criteria

- 1. Female, >18 years of age, with the clinical diagnosis of overactive bladder (based on the current ICS definition<sup>2</sup>).
- 2. Failure of behavioral measures and pharmacologic therapy to adequately control overactive bladder symptoms.
- 3. Baseline patient perception of bladder condition score of 2 or higher.

#### Exclusion criteria

- 1. Current or previous percutaneous or sacral neuromodulation therapy
- 2. Stress predominant urinary incontinence

- 3. Newly added bladder medication or dose change with the last 2 months (Tamsulosin, Silodosin, Alfuzosin, Terazosin, Baclofen, Diazepam, amitriptyline, imipramine, DDAVP, tolterodine, oxybutynin, fesoterodine, darifenacin, solifenacin, trospium, mirabegron)
- 4. Intravesical botulinum toxin use within the last 1 year
- 5. Implanted pacemaker or defibrillator
- 6. History of epilepsy
- 7. Unable or unwilling to commit to study treatment schedule
- 8. Pregnant, or possible pregnancy planned for the duration of the study period
- 9. Active skin disease of the lower legs (dermatitis, cellulitis, eczema, trauma)
- 10. Documented allergy to patch electrodes or their adhesive
- 11. Abnormal sensory function of the lower limb
- 12. Metallic implant within the lower limb

Intervention: Transcutaneous electrical nerve stimulation is a safe and effective therapy that has been used by physicians and other health professionals for a variety of conditions such as pain and muscle rehabilitation<sup>26,27</sup>. We will use the EV-906 Digital TENS machine (from Everyway Medical Instruments Co Ltd, Health Canada License #73631). Two adhesive patch electrodes will be applied to one of the patient's lower limb, and the location used will be based on their treatment assignment (active treatment versus sham). The initial treatment will be carried out in the clinic under the supervision of the investigating physician, with training provided for the patient on proper use of the device by the study nurse. The remaining treatments will be detailed on a calendar for the patient, with telephone contact every 2-3 weeks with research staff to assess compliance. When undergoing active treatment, patients will have the electrodes applied posterior to the medial malleolus, and 5-10 cm above the medial malleolus of the same leg, just behind the medial tibial edge. As per previous studies involving transcutaneous posterior tibial nerve stimulation<sup>25,28,29</sup> and similar to percutaneous tibial nerve stimulation<sup>23</sup>, we will use the bipolar stimulation setting, with a frequency of 10 Hz, 200ms pulse, and the amplitude will be titrated up to patient's maximum nonpainful tolerance (between 0.5-10mA). For patients undergoing sham treatment, they will have the patch electrodes placed on the lateral side of the lower limb, and told to keep the current setting stable at 1mA. This will prevent any meaningful stimulation of the tibial nerve, while still delivering a slight tingling sensation to simulate active treatment.

Primary outcome measure: The patient perception of bladder condition (PPBC) is a commonly used measure for global response in overactive bladder studies. It is an ordinal scale from 0-5 (Appendix 3). It is a valid, reliable and responsive single question asking the patient to select the degree of problems associated with their bladder condition<sup>30</sup>. Patients will be categorized as responders (score improvement by 2 points between screening visit 1 and end of study visit 3) or nonresponders.

#### Secondary outcome measures:

1. OAB related quality of life (OAB-q SF) Valid, reliable, and responsive tool for assessing symptom bother and OAB related quality of life<sup>31</sup>.

- 2. 3-day voiding diary parameters (daily voiding frequency, functional bladder capacity, mean voided volume, longest time between voids, nocturia, number of urgency incontinence episodes). This is a valid and reliable measure of urinary symptoms<sup>32</sup>.
- 3. Quantification of urinary incontinence with 24hr pad weights. This is stable, reliable and responsive measure of the degree of urinary incontinence<sup>33,34</sup>.
- 4. Physician assessment of benefit will be completed based on a standard clinical history at study visit 3 (end of study), and graded on a 7 point global response assessment.

#### Data Analysis and Sample Size

Analysis of our primary outcome will be an intention to treat analysis (using the chi squared test) based on the proportion of patients classified as a responder using the change in the patient perception of bladder condition. A secondary analysis, based on a per protocol analysis (for efficacy) will be performed for patients who completed at least 80% of the treatment sessions for at least 20 min each (determined from patient completed treatment diary, and electronic usage log in the TENS device). Secondary endpoints will be analyzed as appropriate using the students t-test or chi squared test. All data analysis will be carried out using SAS 9.2.

Using previous percutaneous tibial nerve stimulation studies as a guide<sup>23</sup>, we estimate 20% of sham patients and 60% of actively treated patients will be responders. Using the Chi-square test, a two-sided alpha of 0.05, and 80% power, 27 patients per group will be required. Our final sample size, adjusting for a 10% dropout rate, is 60 (30 per group). Our sample size calculation is based on our intention to treat analysis.

#### References

- 1. Welk B, Morrow S, Madarasz W, Baverstock R, Macnab J, Sequeira K. The validity and reliability of the neurogenic bladder symptom score. *J Urol.* 2014;192(2):452-457. doi:10.1016/j.juro.2014.01.027.
- 2. Haylen BT, De Ridder D, Freeman RM, et al. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. *Neurourol Urodyn*. 2010;29(1):4-20. doi:10.1002/nau.20798.
- 3. Stewart WF, Van Rooyen JB, Cundiff GW, et al. Prevalence and burden of overactive bladder in the United States. *World J Urol.* 2003;20(6):327-336. doi:10.1007/s00345-002-0301-4.
- 4. Hartmann KE, McPheeters ML, Biller DH, et al. Treatment of overactive bladder in women. *Evid Rep Technol Assess (Full Rep)*. 2009;(187):1-120, v.
- 5. GARNETT S, Abrams P. The natural history of the overactive bladder and detrusor overactivity. A review of the evidence regarding the long-term outcome of the overactive bladder. *Journal of Urology*. 2003;169(3):843-848. doi:10.1097/01.ju.0000050305.05345.40.
- 6. Abrams P, Kelleher CJ, Kerr LA, Rogers RG. Overactive bladder significantly affects quality of life. *Am J Manag Care*. 2000;6(11 Suppl):S580-S590.
- 7. Tubaro A. Defining overactive bladder: epidemiology and burden of disease. *Urology*. 2004;64(6 Suppl 1):2-6. doi:10.1016/j.urology.2004.10.047.

- 8. Gormley EA, Lightner DJ, Faraday M, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment. *J Urol*. 2015;193(5):1572-1580. doi:10.1016/j.juro.2015.01.087.
- 9. Chapple CR, Khullar V, Gabriel Z, Muston D, Bitoun CE, Weinstein D. The effects of antimuscarinic treatments in overactive bladder: an update of a systematic review and meta-analysis. *European Urology*. 2008;54(3):543-562. doi:10.1016/j.eururo.2008.06.047.
- 10. Tune LE. Anticholinergic effects of medication in elderly patients. *J Clin Psychiatry*. 2001;62 Suppl 21:11-14.
- 11. Sexton CC, Notte SM, Maroulis C, et al. Persistence and adherence in the treatment of overactive bladder syndrome with anticholinergic therapy: a systematic review of the literature. *Int J Clin Pract*. 2011;65(5):567-585. doi:10.1111/j.1742-1241.2010.02626.x.
- 12. Veenboer PW, Bosch JLHR. Long-Term Adherence to Antimuscarinic Therapy in Everyday Practice: A Systematic Review. *Journal of Urology*. 2014;191(4):1003-1008. doi:10.1016/j.juro.2013.10.046.
- 13. Benner JS, Nichol MB, Rovner ES, et al. Patient-reported reasons for discontinuing overactive bladder medication. *BJU Int.* 2010;105(9):1276-1282. doi:10.1111/j.1464-410X.2009.09036.x.
- 14. Andersson K-E.  $\beta$ 3-receptor agonists for overactive bladder--new frontier or more of the same? *Curr Urol Rep.* 2013;14(5):435-441. doi:10.1007/s11934-013-0335-8.
- 15. Oerlemans DJAJ, van Kerrebroeck PEV. Sacral nerve stimulation for neuromodulation of the lower urinary tract. *Neurourol Urodyn*. 2008;27(1):28-33. doi:10.1002/nau.20459.
- 16. Tai C, Chen M, Shen B, Wang J, Roppolo JR, de Groat WC. Irritation induced bladder overactivity is suppressed by tibial nerve stimulation in cats. *J Urol.* 2011;186(1):326-330. doi:10.1016/j.juro.2011.04.023.
- 17. Chang CJ, Huang ST, Hsu K, Lin A, Stoller ML, Lue TF. Electroacupuncture decreases c-fos expression in the spinal cord induced by noxious stimulation of the rat bladder. *Journal of Urology*. 1998;160(6 Pt 1):2274-2279.
- 18. Finazzi-Agrò E, Petta F, Sciobica F, Pasqualetti P, Musco S, Bove P. Percutaneous tibial nerve stimulation effects on detrusor overactivity incontinence are not due to a placebo effect: a randomized, double-blind, placebo controlled trial. *J Urol.* 2010;184(5):2001-2006. doi:10.1016/j.juro.2010.06.113.
- 19. Vandoninck V, van Balken MR, Finazzi-Agrò E, et al. Percutaneous tibial nerve stimulation in the treatment of overactive bladder: urodynamic data. *Neurourol Urodyn.* 2003;22(3):227-232. doi:10.1002/nau.10111.
- 20. Gaziev G, Topazio L, Iacovelli V, et al. Percutaneous Tibial Nerve Stimulation (PTNS) efficacy in the treatment of lower urinary tract dysfunctions: a systematic review. *BMC Urol*. 2013;13:61. doi:10.1186/1471-2490-13-61.
- 21. Peters KM, Carrico DJ, Wooldridge LS, Miller CJ, Macdiarmid SA. Percutaneous tibial nerve stimulation for the long-term treatment of overactive bladder: 3-year results of the STEP study. *J Urol.* 2013;189(6):2194-2201. doi:10.1016/j.juro.2012.11.175.

- 22. Martinson M, MacDiarmid S, Black E. Cost of neuromodulation therapies for overactive bladder: percutaneous tibial nerve stimulation versus sacral nerve stimulation. *J Urol.* 2013;189(1):210-216. doi:10.1016/j.juro.2012.08.085.
- 23. Peters KM, Carrico DJ, Perez-Marrero RA, et al. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. *J Urol.* 2010;183(4):1438-1443. doi:10.1016/j.juro.2009.12.036.
- 24. van der PAL F, van Balken MR, Heesakkers JPFA, Debruyne FMJ, Bemelmans BLH. Percutaneous tibial nerve stimulation in the treatment of refractory overactive bladder syndrome: is maintenance treatment necessary? *BJU Int.* 2006;97(3):547-550. doi:10.1111/j.1464-410X.2006.06055.x.
- 25. Ammi M, Chautard D, Brassart E, Culty T, Azzouzi A-R, Bigot P. Transcutaneous posterior tibial nerve stimulation: evaluation of a therapeutic option in the management of anticholinergic refractory overactive bladder. *Int Urogynecol J.* 2014;25(8):1065-1069. doi:10.1007/s00192-014-2359-0.
- 26. Johnson MI. Transcutaneous Electrical Nerve Stimulation (TENS). Oxford University Press; 2014.
- 27. Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. *J Pain*. 2003;4(3):109-121.
- 28. Amarenco G, ISMAEL SS, Even-Schneider A, et al. Urodynamic effect of acute transcutaneous posterior tibial nerve stimulation in overactive bladder. *Journal of Urology*. 2003;169(6):2210-2215. doi:10.1097/01.ju.0000067446.17576.bd.
- 29. De Seze M, Raibaut P, Gallien P, et al. Transcutaneous posterior tibial nerve stimulation for treatment of the overactive bladder syndrome in multiple sclerosis: results of a multicenter prospective study. *Neurourol Urodyn.* 2011;30(3):306-311. doi:10.1002/nau.20958.
- 30. Coyne KS, Matza LS, Kopp Z, Abrams P. The validation of the patient perception of bladder condition (PPBC): a single-item global measure for patients with overactive bladder. *European Urology*. 2006;49(6):1079-1086. doi:10.1016/j.eururo.2006.01.007.
- 31. Coyne KS, Thompson CL, Lai J-S, Sexton CC. An overactive bladder symptom and health-related quality of life short-form: validation of the OAB-q SF. *Neurourol Urodyn*. 2015;34(3):255-263. doi:10.1002/nau.22559.
- 32. Groutz A, Blaivas JG, Chaikin DC, et al. Noninvasive outcome measures of urinary incontinence and lower urinary tract symptoms: a multicenter study of micturition diary and pad tests. *J Urol.* 2000;164(3 Pt 1):698-701.
- 33. Ryhammer AM, Djurhuus JC, Laurberg S. Pad testing in incontinent women: a review. *Int Urogynecol J Pelvic Floor Dysfunct*. 1999;10(2):111-115.
- 34. FLISSER AJ, Figueroa J, Bleustein CB, Panagopoulos G, BLAIVAS JG. Pad test by mail for home evaluation of urinary incontinence. *Neurourol Urodyn.* 2004;23(2):127-129. doi:10.1002/nau.20023.

## **Appendices**

# A randomized trial of transcutaneous posterior tibial nerve stimulation for refractory overactive bladder patients

### Dr Blayne Welk

- $1. \ \ Key\ randomized\ controlled\ trials\ of\ percutaneous\ tibial\ nerve\ stimulation$
- 2. Schedule of visits for study patients
- 3. Patient perception of bladder condition (PPBC)

**Appendix 1.** Randomized controlled trials evaluating percutaneous tibial nerve stimulation.

| Study | Sample | Design | Intervention/Control | Outcome |
|---|---|---|---|---|
| OrBIT <sup>1</sup> | 100 adults<br>with urinary<br>frequency<br>>8/day and<br>OAB | Randomized<br>controlled trial.<br>Intention to treat. | PTNS (Urgent PC): 0.5-0mA,<br>20Hz, unilateral needle<br>electrode, weekly 30 minute<br>sessions x 12 weeks.<br>Control: Tolterodine 4mg OD<br>x 90 days | Intervention: 80% global response assessment moderate or markedly improved Sham: 55% global response assessment moderate or markedly improved. P<0.01 |
| SUmiT <sup>2</sup> | 220 adults<br>with OAB | Randomized<br>controlled clinical<br>trial. Intention to<br>treat. | PTNS (Urgent PC): 0.5-10mA, 20Hz, unilateral needle electrode, weekly 30 minute sessions x 12 weeks. Control: Sham group with identical setup but no active electricity. | Intervention: 55% global response assessment moderate or markedly improved Sham: 21% global response assessment moderate or markedly improved. P<0.001 |
| PTNS versus<br>placebo <sup>3</sup> | 35 women<br>with<br>urodynamic<br>DO and wet<br>OAB | Randomized<br>controlled trial.<br>Intention to treat. | PTNS (Urgent PC): 0.5-10mA, 20Hz, unilateral needle electrode, 30 minute sessions 3x/week x 12 weeks. Control: Sham group with identical setup but no active electricity. | Intervention: 71% global response assessment moderate or markedly improved Sham: 0% global response assessment moderate or markedly improved. P<0.001 |
| PTNS vs<br>Oxybutynin vs<br>Combination for<br>OAB <sup>4</sup> | 70 women<br>with OAB | Randomized<br>controlled trial. | PTNS (Urgent PC): 0.5-0mA, 10Hz, unilateral needle electrode, weekly 30 minute sessions x 12 weeks. Comparator 1: Oxybutynin SR 10mg PO OD x 12 weeks Comparator 2: Both PTNS and Oxybutynin x 12 weeks | Significant reduction<br>among all groups, and no<br>difference between groups<br>based on ICIQ-SF score. |

Peters KM, Macdiarmid SA, Wooldridge LS, et al. Randomized trial of percutaneous tibial nerve stimulation versus extended-release tolterodine: results from the overactive bladder innovative therapy trial. *J Urol.* 2009;182(3):1055– 1061

<sup>2.</sup> Peters KM, Carrico DJ, Perez-Marrero RA, et al. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. *J Urol.* 2010;183(4):1438–1443.

<sup>3.</sup> Finazzi-Agrò E, Petta F, Sciobica F, Pasqualetti P, Musco S, Bove P. Percutaneous tibial nerve stimulation effects on detrusor overactivity incontinence are not due to a placebo effect: a randomized, double-blind, placebo controlled trial. *J Urol.* 2010;184(5):2001–2006.

<sup>4.</sup> Souto SC, Reis LO, Palma T, Palma P, Denardi F. Prospective and randomized comparison of electrical stimulation of the posterior tibial nerve versus oxybutynin versus their combination for treatment of women with overactive bladder syndrome. *World J Urol.* 2014;32(1):179–184.

## Appendix 2. Study schedule.

| STUDY SCHEDULE | Visit 1 Screening | Visit 2<br>Randomization | Telephone<br>Followup | Visit 3 End<br>of study |
|---|---|---|---|---|
| Visit Windows | 1- 4 weeks<br>prior to<br>Randomization | Week 0 | Every 2-3<br>Weeks | 12-13 Weeks |
| Documentation of Consent | X | | | |
| Medical History and Physical Exam | X | | | |
| Inclusion/ Exclusion Criteria Review | X | | | |
| Medication and Health Review | X | | | X |
| Urine Pregnancy Test | X | | | |
| PPBC Questionnaire | X | | X<br>(week 6-7<br>only) | Х |
| OAB-q SF Questionnaire | X | | | X |
| 3 day Voiding diary | Diary Provided | Completed diary<br>returned & new one<br>provided for Visit 3 | | Completed<br>diary<br>returned |
| 24hr Urinary Pad test | Supplies<br>Provided with<br>instruction | Pads Returned &<br>new ones provided<br>for Visit 3 | Pad test<br>done 1-7<br>days prior to<br>visit 3 | Pads<br>Returned |
| Randomization | | X | | |
| Initial 30 minute treatment session in clinic with nurse supervision | | X | | |
| Assessment of treatment masking | | | X<br>(week 2-3<br>only) | |
| Assessment of compliance, review instructions, address any adverse events or questions | | | X | |
| Physician assessment of benefit | | | | X |

**Appendix 3.** Patient perception of bladder condition. Scored 0 (no problems) to 5 (severe problems).

#### (PPBC)

Which of the following statements describes your bladder condition best at the moment? Please mark "X" in one box only.

My bladder condition does not cause me any problems at all.

My bladder condition causes me some very minor problems.

My bladder condition causes me some minor problems.

My bladder condition causes me (some) moderate problems.

My bladder condition causes me severe problems.

My bladder condition causes me many severe problems.